CLINICAL TRIAL: NCT03504475
Title: An Open-Label Randomized, Single-Dose, 2-way Crossover Bioequivalence Study of Paroxetine Hydrochloride 20 mg Tablets and Paxil® Under Fasting Conditions and Under Fed Conditions in Chinese Healthy Volunteers
Brief Title: Bioequivalence Study of Paroxetine Tablets and Paxil® Under Fasting and Fed Conditions in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: Beijing Winsunny Pharmceutical Co.,Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: WS-CP-06-201709-01
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-05

CONDITIONS: Major Depressive Disorder; Obsessive-Compulsive Disorder; Panic Disorder; Social Anxiety Disorder; Generalized Anxiety Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Obsessive-Compulsive Disorder; Panic Disorder; Phobia, Social; Generalized Anxiety Disorder | interventions — Paroxetine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paroxetine Hydrochloride Tablet (Experimental): During the study session, healthy subjects will be administered a single dose of Paroxetine Hydrochloride Tablet 20mg under Fasting and Fed conditions.
  Interventions: Drug: Paroxetine Hydrochloride Tablet 20 mg
- Paxil® (Active Comparator): During the study session, healthy subjects will be administered a single dose of Paxil® 20mg under Fasting and Fed conditions.
  Interventions: Drug: Paxil® 20 mg

INTERVENTIONS:
Drug: Paroxetine Hydrochloride Tablet 20 mg — A generic product manufactured by Beijing Winsunny Pharmaceutical Co., Ltd.
  Arms: Paroxetine Hydrochloride Tablet
Drug: Paxil® 20 mg — Paxil® Tablet 20 mg will be used as a comparator drug for the bioequivalence study, manufactured by GlaxoSmithKline（Distributed by: Apotex Corp.）.
  Other Names: Paroxetine Hydrochloride Tablet 20 mg
  Arms: Paxil®

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of paroxetine hydrochloride 20 mg tablets (test) and Paxil® (reference) administered as 20 mg tablet under fed conditions.

DETAILED DESCRIPTION:
The study design is an Open-Label Randomized, Single-Dose, 2-way Crossover Bioequivalence Study with a washout period of 14 days. During each session, the subjects will be administered a single dose of 20 mg Paroxetine (one Paroxetine Hydrochloride Tablet 20mg or one Paxil® Tablet 20 mg) under Fasting and Fed conditions. Venous blood samples will be collected at pre-dose (0 h), and up to 96 h post dose.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are fully informed and voluntarily consent to participate in this study.
2. Healthy adult volunteers of ≥18 years old and ≤ 65 years old, male or female.
3. Body weight ≥ 50.0 kg for male and 45.0 kg for female , and body mass index (BMI) ranges from 19.0 to 28.0 kg/m2(including).
4. The results of physical examination, vital signs examination, clinical laboratory examination (blood routine, urine routine, blood biochemistry), 12-lead electrocardiogram (ECG), chest radiograph were normal or no clinical significant.

Exclusion Criteria:

1. Allergy or hypersensitivity to paroxetine or components in the formulation, or have clear history of drug allergies, or have been diagnosed with allergic constitution.
2. History of any diseases which could interfere with the clinical safety or the process in vivo of the drug, such as liver, kidney, cardiovascular, tuberculosis, epilepsy, asthma, diabetes or glaucoma disease, especially the endocrine disease, gastrointestinal disease, gastrointestinal surgery, or unresolved gastrointestinal symptoms (such as diarrhea, vomiting).
3. Present of any unstable or recurrent diseases , or diseases that interfere with the process in vivo of the drug.
4. History of drug abuse/dependence, drug-taking, or positive urine drug screen at screening.
5. Significant alcohol abuse within 2 years ( more than two units of alcohol per day, drink at least 14 units of alcohol per week: 1 unit = 285 mL of beer or 120 mL of white spirit or 25 mL of spirit or 100 mL of wine) ,or positive alcohol exhalation test at screening.
6. Smoking within 1 year (more than 5 cigarettes per day), or could not avoid smoking during the study period started from signing the informed consent forms.
7. Use of any medication changed the liver enzyme activity within the 28 days prior to the study.
8. Use of any medication within 14 days prior to the study.
9. With special diet (including grapefruit and/or xanthine, etc.) or vigorous exercise, or other factors that affected the drug absorption/distribution/metabolism/excretion within 14 days prior to the study.
10. Volunteer in any other clinical drug study within 90 days prior to the study.
11. Blood donation or lost more than 200 mL of blood within 90 days prior to the study.
12. History of needlesickness or hematophobia, or cannot tolerate venipuncture.
13. A positive result in hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibodies, a syphilis test, or an human immunodeficiency virus (HIV) test.
14. Have the family fertility plan, unwilling or unable to take effective contraceptive methods to prevent pregnancy from 30 days before the study until 6 months after the end of study.
15. Positive Human chorionic gonadotropin (HCG) results for female, or lactating women.
16. Have special diet, cannot control diet and exercise as requested.
17. Other situations that the researchers considered unsuitable to enroll the subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-06-16 (Actual)

PRIMARY OUTCOMES:
Cmax | Blood samples collected over 96 hour period
  Maximum Observed Concentration (of Paroxetine in Plasma)
AUC(0-∞) | Blood samples collected over 96 hour period
  Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
AUC(0-t) | Blood samples collected over 96 hour period
  Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zhao, PhD, Principal Investigator — Beijing Tongren Hospital
Locations (2):
- China (2):
  - Beijing TongRen Hospital, Beijing, Beijing Municipality
  - Beijing TongRen Hospital, Beijing